CLINICAL TRIAL: NCT06203353
Title: Evaluation of the Diaphragm Tissue Doppler Parameters in Predicting Weaning From Mechanical Ventilation Outcome
Brief Title: Evaluation of the Diaphragm Performance During Weaning From Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of anesthesiology and ICU department, Mongi Slim Hospital
Other Study IDs: Diaphram Tissue Doppler
Record Dates: First submitted 2023-12-28; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Mechanical Ventilation Weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- weaning success: Patients extubated with no need to non invasive ventilatry support during 48 hours
  Interventions: Diagnostic Test: diaphragm ultrasound monitoring
- weaning failure: patients requiring reintubation or non invasive ventilation within 48 hours after extubation
  Interventions: Diagnostic Test: diaphragm ultrasound monitoring

INTERVENTIONS:
Diagnostic Test: diaphragm ultrasound monitoring — Ultrasound measure the diaphragm excursion, thickening fraction and maximal contraction and relaxation velocities

SUMMARY:
Prospective observationnal study, including ICU adult patients with invasive mechanical ventilation for at least 48 hours. Patients are included when performing weaning from mechanical ventilation with pressure support (lowest level of pressure support).

Before separating the patient from the ventilator and performing a T tube spontaneous breathing test, diaphragm ultrasound is performed bilaterally : diaphragm excursion, diaphragm thickening fraction and maximal contraction and relaxation velocities with tissue doppler imaging.

DETAILED DESCRIPTION:
This observationnal study will include patients during weaning from invasive mechanical ventilation: ventilation in pressure support with the lowest level With normal neurological status: glasgow coma scale > 13 Requiring no vasopressor support

conventionnal diaphragm parameters: diaphram excursion and thickening fraction will be collected bilaterally with the tissue doppler measures: maximal contraction and relaxation velocities, immediately before a T Tube test.

Patients will be divided into 2 groups according to their weaning from mechanicla ventilation outcome, and diaphragm ultrasound patterns will be compared between the 2 groups in order to evaluate the performance of tissue doppler in predicting weaning outcome.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation for at least 48 hours

Exclusion Criteria:

* reintubation for extra respiratory failure (neurologic or hemodynamic)
* Patients with chronic repiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing weaning from mechanical ventilation: Pressure support ventilation with the lowest level of support Glasgow coma scale of at least 13 Hemodynamic stability with no vasopressors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
weaning from mechanical ventilation success | Day 2
  no need of non invasive ventilation or reintubation

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided